CLINICAL TRIAL: NCT00569998
Title: An Open-label, Multi-centre, Multi-national, Comparative, Randomised, Cross-over Trial Evaluating Preference as Well as Performance, Acceptance, Handling and Safety of NovoPen™ 4 (MS236) Versus NovoPen 3® in Insulin Treated Diabetic Patients
Brief Title: Comparison of Two Pen Systems in Patients With Diabetes Treated With Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS236-1544
Record Dates: First submitted 2007-12-04; First posted 2007-12-10 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoPen™ 4
Device: NovoPen® 3

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two insulin delivery pens in the everyday life setting of patients with diabetes treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus for at least 12 months
* Adults at least 18 years
* Children/adolescents between 9-18 years
* HbA1c lesser than or equal to 11.0%

Exclusion Criteria:

* Known or suspected alcohol or drug abuse
* Patients who are not able to read the user manual (may wear glasses if needed)
* Hypoglycaemic unawareness as judged by the investigator
* Visual and/or dexterity impairments as judged by the investigator

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2003-08; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of overall pen preference | after 12 weeks of treatment

SECONDARY OUTCOMES:
HbA1c
Adverse device effects
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (21):
- Novo Nordisk Investigational Site, Vienna, Austria
- Germany (6):
  - Novo Nordisk Investigational Site, Cologne
  - Novo Nordisk Investigational Site, Leverkusen
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Völklingen
- Italy (5):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Parma
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Torino
- Netherlands (6):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Heerlen
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Veldhoven
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Sidcup

REFERENCES:
- [Result] Kolaczynski M, Chayer D. NovoPen® 4: perceived as superior in handling and acceptance versus HumaPen® Ergo and OptiPen® Pro in patients and healthcare professionals. Diabetes Technology & Therapeutics 2005; 7 (2): 390
- [Result] Goke B, Gamba S, Erdtsieck RJ, Gilbey S, Schober E, Lytzen L, Kolaczynski M. NovoPen 4 offers superior performance, handling and acceptance compared with NovoPen 3 in insulin-treated diabetes patients. Diabetes Technology and Therapeutics 2005; 7 (2): 379-380
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com